CLINICAL TRIAL: NCT06437834
Title: Increasing Men's Engagement in Preventive Healthcare Through an Enhanced Cocoon Vaccination Strategy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY20240985; UM1TR004528 (NIH)
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Vaccines; Preventive Medicine
Keywords: cocoon vaccination; men's health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaccination Offer only (No Intervention): all male-identifying visitors in the birthing center will receive the offer of influenza and Tdap vaccinations at the bedside only.
- Offer of Bedside Vaccines plus Information (Experimental): All male-identifying visitors in the birthing center at the birthing center will receive an information sheet about vaccinations and preventive healthcare, and will be offered influenza and Tdap vaccinations at bedside in the birthing center.
  Interventions: Other: Information Sheet
- Offer of Bedside Vaccines plus High-touch connection (Experimental): All male-identifying visitors in the birthing center will receive the information sheet, and will be offered influenza and Tdap vaccinations at bedside in the birthing center, as well as a high-touch connection to healthcare navigation supports.
  Interventions: Other: Information Sheet; Other: High-touch connect

INTERVENTIONS:
Other: Information Sheet — Information sheet describing the importance of vaccines and preventive care as well as contact information for patient navigators.
  Arms: Offer of Bedside Vaccines plus High-touch connection; Offer of Bedside Vaccines plus Information
Other: High-touch connect — Engagement with a patient navigator.
  Arms: Offer of Bedside Vaccines plus High-touch connection

SUMMARY:
The goal of this clinical trial is to understand if offering a high touch engagement with healthcare center catered to men and bedside vaccine access in a birthing center increases men's engagement in preventive healthcare. The main questions it aims to answer are:

Does access to vaccinations and overall health education for men lead to increased uptake of vaccines? Does access to vaccinations and overall health education for men lead to increased engagement in overall healthcare of male identifying support persons.

Researchers will compare three arms (one that receives an offer of vaccines at bedside in the birthing clinic, one that receives an information flyer about the importance of preventive care in addition to the offer of vaccines and a third one that receives higher level of engagement from patient liaisons as well as the offer of vaccines at bedside) to see if there is a difference in vaccine uptake and engagement in healthcare.

Outcomes will be measured by aggregate number of men receiving vaccines weekly in each arm and aggregate number of men enrolling in a men's health care center in each arm. Men will also be invited to complete a survey and a portion will be invited to complete and interview.

DETAILED DESCRIPTION:
The goal of this project is to understand whether the combination of vaccination access and connection to services tailored for men improves vaccination rates among men and engagement in healthcare. Additionally, this project aims to understand variations in effectiveness between low-touch and high-touch approaches. To achieve these goals, the project has two specific aims:

Aim 1: Assess the effectiveness of cocoon vaccination interventions on a continuum of minimum to high-touch in terms of vaccination completion and healthcare engagement. After refinement of the intervention materials and study materials based on engagement with community members, representatives of the priority population, interested parties including birthing parents, the initiative will roll out in three randomly timed clusters, one that includes bedside vaccinations, another that includes bedside vaccinations in addition to low-touch informational flyer, and a third that includes bedside vaccinations and high-touch connection to the UH Cutler Center for Men through the Joe Team. Vaccination completion will be assessed utilizing records from the Pharmacy department delivering the vaccinations. Health care engagement will be assessed utilizing records from the UH Cutler Center for Men on enrollment in the center. Male-identifying individuals will also be recruited and enrolled to complete a survey at baseline to assess healthcare engagement.

Aim 2: Examine the factors that impact uptake of vaccination and healthcare engagement after a cocoon vaccination intervention. Factors that impact intervention uptake will be assessed through the survey and semi-structured interviews with a subsample of survey participants. Additionally, contextual factors related to the implementation of the intervention, such as hours of operation for high touch connections/vaccine distribution will be assessed. By understanding the factors that impact intervention uptake, we will assess the barriers and facilitators of this strategy.

Hypothesis. This pilot study will examine whether implementing a cocoon vaccination strategy that provides access to vaccinations and overall health education for men leads to increased uptake of vaccines and engagement in overall healthcare of male identifying support persons. Additionally, it will assess the factors that impact intervention uptake. We anticipate that vaccination rates and engagement with healthcare will be highest among male visitors at the Ahuja Medical Center who receive the vaccination offer at bedside and the high-touch healthcare navigation information relative to those who are only offered offered bedside vaccines only.

ELIGIBILITY:
Inclusion Criteria:

- Adult Partner of birthing person at a birthing center who identifies as male-identifying

Exclusion Criteria:

-Under the age of 18; does not identify as a man.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identifies as Male
Enrollment: 176 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Number of male-identifying individuals who received Influenza Vaccine | Up to 7 weeks
  Aggregate number of influenza vaccinations provided in the birthing center utilizing pharmacy records

SECONDARY OUTCOMES:
Number of male-identifying individuals who received TDap Vaccine | Up to 7 weeks
  Aggregate number of Tdap vaccinations provided in the birthing center utilizing pharmacy records
Number of participant who enrolled in Patient Navigation | Up to 7 weeks
  Enrollment in Men's Health Center that includes patient navigation from records from the Men's Health Center

CONTACTS AND LOCATIONS:
Overall Officials: Randy Vince, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT06437834/ICF_000.pdf